CLINICAL TRIAL: NCT02833467
Title: A Prospective Study of Identifying Genomic Mutations of Multiple Primary Lung Cancers by Circulating Tumor DNA
Brief Title: Identifying Genomic Mutations of Multiple Primary Lung Cancers by Circulating Tumor DNA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: San Valley Biotechnology Incorporated (Unknown)
Responsible Party: Principal Investigator, Chen KeZhong, MD，Thoracic Surgery Service, Peking University People's Hospital
Other Study IDs: PTHO1502
Record Dates: First submitted 2016-07-09; First posted 2016-07-14 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Carcinoma; Non-small-cell Lung Cancer; Thoracic Neoplasms
Keywords: Circulating Tumor DNA; Heterogeneous; Multiple primary lung cancer
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung; Thoracic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh tumor tissue, peripheral blood cells, and plasma samples were collected from each patient.
Oversight: Data Monitoring Committee: No

SUMMARY:
Targeted next generation sequencing (NGS) provides a promising method for diagnostic purposes by enabling the simultaneous detection of multiple gene mutations. This study is to evaluate the feasibility and application value by using NGS into identifying genomic mutations in multiple or multifocal primary lung cancers in cell-tumor DNA (ctDNA) from surgical patients

DETAILED DESCRIPTION:
Tumor samples originating from clinically considered multiple or multifocal primary lung cancer patients were available for mutational analysis. DNA and RNA were extracted from fresh tumor tissue or formalin-fixed, paraffin-embedded (FFPE) tissue. A series of cancer-related genomic alterations including single nucleotide variations (SNVs), short insertions and deletions (InDels), copy number variations (CNVs) and gene rearrangements were identified by a comprehensive NGS Panal . High frequency mutations were also identified in blood sample by droplet digital polymerase chain reaction(ddPCR).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have given written informed consent
* Histopathologically confirmed NSCLC
* Considered multiple or multifocal primary lung cancer by clinical criteria

Exclusion Criteria:

* Malignant tumor history within the past 5 years
* Patients who received any treatment prior to resection
* Insufficient tumor tissue or blood sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple or multifocal primary lung cancer patients who underwent surgery
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-01; Primary Completion 2020-01 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
The detection rate of cancer related genes in multiple primary lung cancer patients by targeted next generation sequencing | 18 months

SECONDARY OUTCOMES:
The concordant and discordant frequency of genomic results between tumor tissue and circulating tumor DNA in multiple primary lung cancer patients | 18 months
The relationship between disease free survival and genomic results in multiple primary lung cancer patients | 5 years
The relationship between overall survival and genomic results in multiple primary lung cancer patients | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kezhong Chen, M.D., Principal Investigator — Peking University People's Hospital; Jun Wang, M.D., Study Chair — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: Undecided